CLINICAL TRIAL: NCT01809288
Title: Identifying Risk for Diabetes and Heart Disease in Women: A Study of African-American, African and White Federal Employees and Contractors
Brief Title: Identifying Risk for Diabetes and Heart Disease in Women
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 130090; 13-DK-0090
Record Dates: First submitted 2013-03-09; First posted 2013-03-12 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-08-21

CONDITIONS: Obesity; Insulin Resistance; Triglycerides; Diabetes
Keywords: Women; Diet; Obesity; African; Physical Activity; Natural History
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Healthy African, African-American, and white women between 30 and 65 years of age who are federal employees or contractors.

SUMMARY:
Background:

- Rates of diabetes and heart disease in women are increasing. Early recognition of risk could help women live longer and healthier lives. Race and ethnicity may affect the best kinds of tests to use to screen for these conditions. Researchers want to compare risk factors for diabetes and heart disease in African, African-American, and white women. Doing so may help identify the most effective screening test for each group. This study will look at healthy African, African-American, and white women who are federal employees and contractors.

Objectives:

- To study risk factors for diabetes and heart disease in African, African-American, and white women.

Eligibility:

* Healthy African, African-American, and white women between 30 and 65 years of age who are federal employees or contractors.
* For this study, African women must be born in Africa and have immigrated to the United States, and report that both parents are Africans. African-American women must self-identify as African-Americans, born in the United States, and have parents who both self-identify as African-American born in the United States. White women must self-identify as white and have parents who also self-identify as white.

Design:

* Participants will have four visits to study their risk factors for diabetes and heart disease.
* The first visit is a screening visit. Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected. They will also have an EKG test. Participants will also be shown how to fill out a 3-Day Food Record and wear an activity monitor called an accelerometer. The food record will keep track of how much participants eat for 3 consecutive days, including 1 non-working day. The accelerometer device will be worn for 3 days to monitor movement.
* At the second visit, participants will have blood tests, an oral glucose tolerance test, and body fat measurements. They will also fill out questionnaires, review the food record, and have two imaging studies.
* At the third visit, participants will have a longer glucose tolerance test. During the test, participants will receive both glucose and insulin and blood samples will be collected over several hours. Participants will receive lunch at the clinical center after the test.
* At the fourth visit, participants will have a meal test. They will fast for 12 hours before the test. Participants will eat a specific meal and have blood samples taken during and after they eat.
* Participants will discuss the results of these tests with the study doctors.

DETAILED DESCRIPTION:
African-American women experience disproportionately high rates of conditions related to insulin resistance, specifically type 2 diabetes (T2D) and cardiovascular disease (CVD). In Africa, T2D and CVD have also become leading causes of death for women. Early recognition of risk and the implementation of preventive measures could improve both quality of life and longevity as well as decrease health care expenditures. However, screening tests for the early detection of T2D and CVD were developed several decades ago in large studies with mostly white participants. Emerging evidence suggests that there are racial differences in the ability and importance of various risk factors to predict the development of diabetes and CVD. Consequently tests used to screen for T2D and CVD are often not effective in women of African descent. Thus, women of African descent lose the opportunity and benefit of early intervention.

Designing tests to determine risk for T2D and CVD in women of African descent requires an appreciation of why current tests do not work. Screening tests to detect risk for T2D and CVD usually rely on the observation that insulin resistance is associated with increased hepatic fat, high fasting glucose and high triglyceride (TG) levels. However, while insulin-resistant white women usually have high liver fat, high fasting glucose and high TG levels, insulin-resistant African-American women often have normal TG levels, normal fasting glucose and low hepatic fat. Therefore, these tests routinely fail to detect risk in African-American women.

The relationship between TG levels to insulin resistance, hepatic glucose production and liver fat has not been studied in African women. To improve diagnosis, we propose a study of race differences in TG levels, fasting glucose levels and hepatic fat comparing 3 groups of women who are federal employees or contractors: African-American African (born in subSaharan Africa and immigrated to the United States) and white. This design ensures all enrollees will have health insurance, a similar work environment and a comparable distribution of position (i.e. scientific, administrative, support). Analyses to detect differences in diet, physical activity and other psychosocial factors will be undertaken.

There will be 4 outpatient visits for 360 non-diabetic women (120 African-American, 120 African and 120 white, aged 25 to 65 years, BMI 20 to 45 kg/m2) enrolled. At Visit 1, a medical history, physical exam and screening labs will be done. Participants will record food intake and monitor physical activity wear an activity monirot (accelerometer) during a 7-day period between visits. At Visit 2 an oral glucose tolerance test will be performed. Studies to examine body fat content and distribution will also be done. At Visit 3, insulin resistance will be measured with an intravenous glucose tolerance test. At Visit 4, breakfast will be eaten with blood samples taken before and after the meal.

In addition to the 4 outpatient visits described, there will be an optional overnight stay the evening before visit 3 for 60 women (30 African descent and 30 white). The purpose of this smaller study is to determine if race differences in the production of glucose by the liver contribute to race differences in fasting glucose levels. Eligible women will be in good health, between 25 and 50 years of age and have a BMI 25-45kg/m2.

This study will be the first time (a) TG levels in African immigrants are compared to African-American and white women (b) hepatic glucose production is assessed by race, and (c) the relationship of TG to insulin resistance, liver fat, body fat distribution, diet, physical activity and psychosocial factors are examined in these 3 groups of women under similar metabolic and economic conditions. While failure of screening tests means a lost opportunity for early intervention, effective screening tests can change outcomes, improve lives and minimize health care expenditures. This protocol is building a foundation on which effective screening tests for diabetes and heart disease can be built.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PRIMARY PROTOCOL:
* African, African-American and White Women
* Healthy Volunteers
* Age between 25 and 65 years
* BMI between 20 and 45 kg/m(2)
* Federal Employees-Intramural or Extramural or Contractor

INCLUSION CRITERIA FOR NESTED INPATIENT STUDY

Same as primary outpatient protocol except:

* Age restricted to 25 to 50 years
* BMI restricted to 25 and 45 kg/m2
* Premenopausal status

EXCLUSION CRITERIA:

* Pregnancy
* Medications or Medical Conditions which affect parameters under investigation

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women-Federal Employees and Contractors@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2013-09-26 (Actual); Primary Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Determine if there are differences in African, African-American and white women in the relationship between triglyceride levels, (a frequently used screening test for diabetes and heart disease) glucose tolerance status and insulin resistance. | 2-6 weeks
  Triglyceride concentration and insulin resistance measured by the frequently sampled intravenous glucose tolerance test.

SECONDARY OUTCOMES:
Determine if there are race or ethnic differences in the pancreatic secretion of insulin relative to the degree of insulin resistance. | 2-6 weeks
  Insulin secretion measured by frequently sampled intravenous glucose tolerance test.

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie T Chung, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Chung ST, Cravalho CKL, Meyers AG, Courville AB, Yang S, Matthan NR, Mabundo L, Sampson M, Ouwerkerk R, Gharib AM, Lichtenstein AH, Remaley AT, Sumner AE. Triglyceride Paradox Is Related to Lipoprotein Size, Visceral Adiposity and Stearoyl-CoA Desaturase Activity in Black Versus White Women. Circ Res. 2020 Jan 3;126(1):94-108. doi: 10.1161/CIRCRESAHA.119.315701. Epub 2019 Oct 18. PMID 31623522
- [Derived] Chung ST, Galvan-De La Cruz M, Aldana PC, Mabundo LS, DuBose CW, Onuzuruike AU, Walter M, Gharib AM, Courville AB, Sherman AS, Sumner AE. Postprandial Insulin Response and Clearance Among Black and White Women: The Federal Women's Study. J Clin Endocrinol Metab. 2019 Jan 1;104(1):181-192. doi: 10.1210/jc.2018-01032. PMID 30260396
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-DK-0090.html